CLINICAL TRIAL: NCT00525434
Title: Evaluation of Safety and Efficacy of Using Seraffix LTB - (Laser Tissue Bonding) System for Excisional Biopsy Wounds Closure
Brief Title: Evaluation of Safety and Efficacy of Using Seraffix LTB - System for Excisional Biopsy Wounds Closure
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: sponsor has decide to pospone this study
Sponsor: Seraffix (Industry)
Responsible Party: Dr. Hanna Levy, Clinical Study Consultant, Seraffix
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SF-EB -01
Record Dates: First submitted 2007-09-04; First posted 2007-09-05 (Estimated); Last update posted 2011-06-09 (Estimated); Status verified 2008-05

CONDITIONS: Dehiscence, Surgical Wound
Keywords: Laser bonding soft tissue albumin
MeSH Terms: conditions — Surgical Wound Dehiscence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Device: Seraffix LTB

INTERVENTIONS:
Device: Seraffix LTB — wounds closure by using laser and albumin

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of using Seraffix LTB system for excisional biopsy wounds closure

DETAILED DESCRIPTION:
Excisional biopsy of the skin is a biopsy in which an entire lesion is removed. An excisional biopsy is in contrast to an incisional biopsy in which only a sample of tissue is cut into and removed. It is most frequently done to diagnose a skin growth such as a mole, or cancer of the skin.

The most common method of wound closure of skin excisions is interrupted nonabsorbable sutures. The sutures should be removed as soon as adequate intrinsic bonding strength is sufficient, depending mostly on the specific body region (from 5-7 days for the face and up to 12-14 days for trunk and extremities).

Laser energy, also known as laser welding, has been used on limited basis as an alternative to traditional wound closure method. There have been two fundamental approaches to laser assisted bonding of tissues:

1. Laser welding-heating the approximated edges of cuts in tissues by a laser beam;
2. Laser soldering- applying a biological solder onto the approximated edges and heating the solder (and the underlying tissue).

Seraffix has developed the Seraffix LTB (Laser Tissue Bonding) System - a laser system for soft tissue bonding. This innovative system includes features that make laser soldering suitable for clinical use. The Seraffix system is composed of CO2 laser device, propriety grip device (Clamps) and soldering agent (Human Albumin).

ELIGIBILITY:
Inclusion Criteria:

1. Male/Female age 18-60.
2. Subject is scheduled for excisional biopsy surgery.
3. Subject able to comprehend and give informed consent for participation in this study.
4. Signed informed consent form.

Exclusion Criteria:

1. Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months prior to screening.
2. Acute infection requiring intravenous antibiotics at the time of screening.
3. Bleeding, coagulation and or clotting disorders.
4. Diabetes mellitus: IDDM or NIDDM.
5. HIV positive or any other immunosuppressive disorder.
6. Renal failure (Serum creatinine >2.0 mg/dl).
7. Inflammatory and or allergic diseases or condition of the skin: Psoriasis, Eczema or dermatitis.
8. Any concomitant infection - viral or bacterial.
9. Drug abuse.
10. Use of steroids.
11. Infection / abscess / pain in treatment target area.
12. Pregnancy or lactating.
13. History of keloid scarring.
14. Use of aspirin or antioxidants
15. Subject is suffering extreme general weakness.
16. Subject objects to the study protocol.
17. Known cognitive or psychiatric disorder
18. Concurrent participation in any other clinical study.
19. Physician objection.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2008-11; Primary Completion 2009-07 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Primary study endpoint will be to establish the safety of using the Seraffix System for excisional biopsy wounds closure. Safety will be established by paucity of serious adverse events and adverse events. | 3 months

SECONDARY OUTCOMES:
1. Re-intervention: A subject is scored a success (1) if he had No Re-intervention by 3 months; otherwise he is scored a failure (0). 2. Wound dehiscence of at least 50% of wound length: | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Yehuda Ullmann, Dr., Principal Investigator — RAMBAM Medical Center, Haifa Israel
Locations (1):
- RAMBAM Medical center, Haifa, Israel